CLINICAL TRIAL: NCT07168668
Title: Exploring Clinical Efficacy of Partial Immune-boost TACE in unrEseCTable HCC Patients Under Systemic Treatment (EXEPECT Trial)
Brief Title: Partial Immune-boost TACE in unrEseCTable HCC Patients Under Systemic Treatment
Acronym: EXEPECT
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202500378B0; NSTC 112-2314-B-182A-016-MY3 (Other Grant/Funding Number: National Science Council, Taiwan)
Record Dates: First submitted 2025-09-03; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: HCC; Tace; Immunotherapy
Keywords: hepatocelluar carcinoma; transarterial chemoembolization; immunotherapy
MeSH Terms: interventions — durvalumab; tremelimumab; atezolizumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- partial TACE with systemic treatment (Experimental): partial TACE
  Interventions: Procedure: Transarterial chemoembolization; Drug: durvalumab and tremelimumab

INTERVENTIONS:
Procedure: Transarterial chemoembolization — 1. Targeting 1-3 prognostically relevant tumor nodules.
  2. Administration of anti-cancer drugs (doxorubicin 20 mg in each section of TACE).
  3. Embolization with Drug-Eluting Beads (doxorubicin 20 mg loaded Hepasphere 20 mg of TACE)
  4. Embolization was done when there was a slight decrease in blood flow for each tumor feeder.
Drug: durvalumab and tremelimumab — Combine TACE with immunotherapy
  Other Names: Atezolizumab & Bevacizumab

SUMMARY:
Study Objectives： Atezolizumab (anti-programmed death-ligand 1; anti-PD-L1) combined with bevacizumab (anti-vascular endothelial growth factor; anti-VEGF) or Durvalumab (anti-programmed death-ligand 1; anti-PD-L1) combined with tremelimumab (anti-cytotoxic T-lymphocyte-associated protein 4; anti-CTLA4) have recently been established as a standard first-line systemic treatment for unresectable hepatocellular carcinoma (HCC). However, its objective response rate (ORR) is only less than 27% (1, 2), and the majority of patients died of HCC progression and liver failure. Therefore, there is an urgent need to develop a novel combination treatment strategy to overcome resistance to immunotherapy and improve patient outcomes.

Transarterial chemoembolization (TACE) remains the standard treatment for patients with intermediate-stage hepatocellular carcinoma (HCC) (3, 4). However, in our previous retrospective study (5-7), the investigators consistently observed that this combination not only improves therapeutic responses but also significantly prolongs patient survival. The tumor necrosis caused by TACE may enhance the efficacy of systemic therapies by promoting the release of neoantigens, thereby stimulating immune responses (8-14). This concept has been substantiated in two recent trials involving intermediate-stage HCC (15, 16), where the addition of immune checkpoint inhibitors to TACE resulted in improved clinical outcomes. Nevertheless, this promising approach has yet to replace the decades-old standard treatment protocols, underscoring the need for further proof-of-concept studies.

Both immunotherapy (atezolizumab/bevacizumab or durvalumab/tremelimumab) and transarterial chemoembolization (TACE) are approved treatment modalities for unresectable hepatocellular carcinoma (HCC) by the U.S. and Taiwan Food and Drug Administration (FDA). This phase II non-randomized trial is designed to prospectively evaluate the therapeutic efficacy, safety, and immunological responses in patients with unresectable HCC treated with a combination of immunotherapy and TACE. A particular focus of this study is to explore the potential immune-boosting effects of TACE, including its ability to enhance antigen presentation and stimulate anti-tumor immune responses.

ELIGIBILITY:
inclusion criteria:

1. Participants must have diagnosis of HCC that is deemed unsuitable for surgical resection or transplant. Participants may have multiple lesions with a total maximal tumor dimension of < 20 cm, and no one lesion > 15 cm. Diagnosis should be confirmed by at least 1 criterion listed below:

   Histologically or cytologically proven diagnosis of HCC. Typical arterial enhancement and delayed washout on multiphasic CT or MRI.
2. Age ≥18 years at the time of signing informed consent document.
3. ECOG performance status 0-1.
4. Barcelona Clinic Liver Cancer (BCLC) stages B or C.
5. Child-Pugh score 5-6 liver function within 28 days of study registration.
6. Documented virology status of hepatitis B virus (HBV), as confirmed by screening HBV serology test.
7. Documented virology status of hepatitis C virus (HCV), as confirmed by screening HCV serology test.
8. Ability to understand and the willingness to sign a written informed consent document
9. Adequate bone marrow, liver, and renal function within 4 weeks before study registration

   * Hemoglobin ≥ 9.0 g/dL
   * Absolute neutrophil count (ANC) ≥ 1,000/mm3
   * Platelet count ≥ 50,000/μL
   * Total bilirubin < 2.5 mg/dL
   * Serum albumin >2.8 g/dL
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 × upper limit of normal (ULN)
   * Prothrombin time ≤ 6 seconds prolonged
   * Serum creatinine ≤ 1.5 mg/dL

Exclusion Criteria:

1. Prior invasive malignancy unless disease free for a minimum of 2 years
2. Prior radiotherapy to the region of the liver that would result in overlap of embolization fields
3. Prior selective internal radiotherapy/hepatic arterial yttrium therapy, at any time
4. Untreated active hepatitis B or hepatitis C
5. Moderate to severe or intractable ascites
6. Untreated or incomplete treated esophageal or gastric varices
7. Severe, active co-morbidity, defined as follows:

   * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months prior to registration
   * Myocardial infarction within the last 6 months prior to study entry
   * Acute bacterial or fungal infection requiring intravenous antibiotics within 28 days prior to study entry
   * A bleeding episode within 6 months prior to study entry due to any cause. o Thrombolytic therapy within 28 days prior to study entry.
   * Known bleeding or clotting disorder.
   * Uncontrolled psychotic disorder
8. Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception
9. Prior solid organ transplantation.
10. Prior or active autoimmune disease (AID) including autoimmune hepatitis, inflammatory bowel disease, myasthenia gravis, systemic lupus erythematosus, rheumatoid arthritis, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjogren's syndrome, Guillain-Barre syndrome, and multiple sclerosis.
11. Prior or active thrombotic or bleeding disorders, hemoptysis, cerebral vascular accident, significant cardiac disease (ischemic or congestive heart failure), or gastrointestinal perforation.
12. Known HIV infection.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 90 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2028-05-30 (Estimated); Study Completion 2028-05-30 (Estimated)

PRIMARY OUTCOMES:
PFS | From enrollment to the end of treatment at 12 months
  PFS 12 month

SECONDARY OUTCOMES:
ORR | 12 months
  Best ORR
OS | OS 3 years
  OS 3 years
DOR | Up to 3 years
  Duration of response
The function of innate CD8+ T cells | Up to 3 years
  Evaluate innate-like CD8⁺ T-cell function using participants' peripheral blood mononuclear cells (PBMCs).

IPD SHARING:
Plan to Share IPD: Undecided